CLINICAL TRIAL: NCT06960538
Title: PRIORITY (Enpowering Progression Risk of Cerebral Amyloid Angiopathy)
Brief Title: Enpowering Progression Risk of Cerebral Amyloid Angiopathy
Acronym: PRIORITY
Status: Recruiting | Type: Observational
Sponsor: Fondazione I.R.C.C.S. Istituto Neurologico Carlo Besta (Other)
Responsible Party: Sponsor
Other Study IDs: PRIORITY
Record Dates: First submitted 2025-04-02; First posted 2025-05-07 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-04

CONDITIONS: Cerebral Amyloid Angiopathy; CAA - Cerebral Amyloid Angiopathy
Keywords: Cerebral Amyloid Angiopathy; CAA; plasma biomarkers; cerebrospinal fluid biomarkers
MeSH Terms: conditions — Cerebral Amyloid Angiopathy; Cerebral Amyloid Angiopathy, Familial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Each patient will undergo CSF collection at baseline (T0) and blood sampling at T0, T1, and T2. CSF is collected via lumbar puncture, processed according to international guidelines, centrifuged, aliquoted, and stored at -80 °C. Blood plasma is isolated using Ficoll gradient centrifugation and similarly stored. CSF biomarkers (Aβ42, Aβ40, t-Tau, p-Tau) are measured via LUMIPULSE G assays (Fujirebio); plasma markers (Aβ42, Aβ40, t-Tau, NfL, GFAP) via ELISA or SIMOA (Quanterix). Untargeted lipidomic profiling (qTOF) of CSF and plasma includes sterols, glycerolipids, phospholipids, sphingolipids, fatty acids, and ether lipids. All patients undergo apoE genotyping; those with family history of CAA, ICH, or cognitive decline are screened for APP, TTR, and PSEN1 variants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Cerebral amyloid angiopathy (CAA) is a microangiopathy characterized by the progressive deposition of β-amyloid in cerebral vessel walls, contributing to intracerebral hemorrhages, cognitive decline, and other clinical manifestations. Despite recent advances in diagnosis and understanding, many pathogenic, prognostic, and therapeutic aspects remain unclear.

Study Objective:

PRIORITY is a prospective observational study aimed at identifying clinical, neuroradiological, and biochemical biomarkers that could improve early diagnosis, risk stratification, and the identification of personalized therapeutic targets for CAA.

DETAILED DESCRIPTION:
PRIORITY is a prospective, single-center observational study conducted at the Fondazione IRCCS Istituto Neurologico Carlo Besta in Milan. It will consecutively enroll patients over 18 years of age with possible or probable cerebral amyloid angiopathy (CAA), symptomatic or asymptomatic, with or without histological confirmation. Diagnosis will follow the updated Boston criteria 2.0, and a brain MRI is mandatory for inclusion.

The study duration is 36 months, with clinical and neuroimaging assessments at baseline (T0), 12 months (T1), and 24 months (T2). CSF analysis will be performed at T0; plasma biomarkers (via ELISA and SIMOA) will be assessed at all time points. Lipid profiles will be analyzed using mass spectrometry with both untargeted and targeted lipidomic approaches (e.g., sphingolipidomics).

The comprehensive clinical and biological dataset will be used to develop a machine learning-based predictive model to support diagnostic, prognostic, and therapeutic decision-making in CAAThe study duration is 36 months, with clinical and neuroimaging assessments at baseline (T0), 12 months (T1), and 24 months (T2). CSF analysis will be performed at T0; plasma biomarkers (via ELISA and SIMOA) will be assessed at all time points. Lipid profiles will be analyzed using mass spectrometry with both untargeted and targeted lipidomic approaches (e.g., sphingolipidomics).

ELIGIBILITY:
Inclusion Criteria:

* patients of either sex over 18 years of age;
* patients with possible and probable symptomatic or asymptomatic CAA with or without histological demonstration (modified Boston criteria);
* patients who have had at least one brain MRI.

Exclusion Criteria:

* patients who have contraindications to undergoing brain MRI (e.g., pacemaker, incompatible mechanical valves, claustrophobia);
* patients who have contraindications to or refuse to undergo lumbar puncture;
* patients who are unable to provide informed consent for the study due to aphasic or cognitive impairment;
* patients who are pregnant or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with possible or probable CAA identified on brain MRI according to modified Boston Neuroradiological Criteria 2.0 regardless of age.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Clinical Progression of CAA | Baseline (T0), 12 months (T1), 24 months (T2).
  Evaluation of the natural progression of cerebral amyloid angiopathy (CAA) through clinical assessments.
  At baseline, clinical data (e.g., history of stroke, a diagnosis of dementia, presence of seizures, gait disturbances, vascular risk factors, prior brain injury/surgery, family history, medications…) recorded in a binary (yes/no) scale, indicating the presence or absence of each condition or risk factor, will be collected for each patient.
  During follow-up, new clinical events (e.g., number of new ICH-intracerebral hemorrhages, number of new ischemic stroke, presence of seizures, presence of TFNEs, cognitive status, death) will be recorded and compared with T0.
Radiological Progression of CAA | Baseline (T0), 12 months (T1), 24 months (T2).
  Evaluation of the natural progression of cerebral amyloid angiopathy (CAA) through neuroimaging markers (MRI).
  MRI assessment at baseline will include T1, T2, FLAIR, T2*, GRE, SWI, and DWI sequences. Imaging will be assessed using STRIVE (Standards for Reporting Vascular Changes on Neuroimaging) criteria, with standardized rating scales for: number of Microbleeds (Microbleed Anatomical Rating Scale - MARS); presence of Lobar ICH- intracerebral hemorrhages; presence of Superficial siderosis; presence of White matter lesions (Fazekas scale: o to 3 scores, where 0 means absence of white matter lesions and 3 large presence of them); presence of Perivascular spaces (CSO-PVS); presence of Cortical microinfarcts; presence of Global cortical atrophy; presence of Subarachnoid haemorrhage.
  Follow-up includes repeated MRI with the same sequences. MRI changes will be evaluated with the same standardized rating scales for progression or appearance of the same parameters evaluated in T0.
Identification of Protein and Lipid Biomarkers | Baseline (T0), 12 months (T1), 24 months (T2).
  Analysis of cerebrospinal fluid and plasma to identify protein (e.g., concentrations in pg/mL of total Tau, p-Tau, Aβ42/Aβ40, NfL, GFAP) and lipid (qTOF-MS) signatures associated with CAA progression.

SECONDARY OUTCOMES:
Cognitive Decline Assessment | Baseline (T0), 12 months (T1), 24 months (T2).
  Longitudinal evaluation of cognitive functions and disability to correlate with disease progression. A neuropsychological evaluation will be performed using the Montreal Cognitive Assessment (MoCA) test, scores range from 0 to 30, with lower scores indicating greater cognitive impairment.
Development of a Predictive Model for Disease Progression | 24 months (T2).
  Development and validation of machine learning models (e.g., Random Forest, Decision Trees) to predict disease progression. Performance metrics include accuracy, sensitivity, specificity, PPV, NPV, and AUC based on integrated clinical, imaging, and biomolecular data.
Hemorrhagic and Non-Hemorrhagic Event Incidence | 24 months (T2)
  Monitoring of symptomatic and asymptomatic cerebral hemorrhages, as well as other vascular events, to determine risk factors.
Therapeutic Target Identification | 24 months (T2)
  Identification of potential molecular targets for future therapeutic interventions based on CSF and plasma biomarker analysis.
Functional assessment | Baseline (T0), 12 months (T1), 24 months (T2)
  Disability will be assessed with the modified Rankin Scale (mRS, scores ranges from 0 - no symptoms - to 6 - death).

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione IRCCS Istituto Neurologico Carlo Besta, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pollaci G, Potenza A, Gorla G, Carrozzini T, Marinoni G, De Toma C, Canavero I, Rifino N, Boncoraglio GB, Difrancesco JC, Damavandi PT, Stanziano M, Erbetta A, Caroppo P, Di Fede G, Catania M, Zulueta A, Parati EA, Bersano A, Gatti L, Storti B. CSF and Plasma Biomarkers in Patients With Iatrogenic Cerebral Amyloid Angiopathy. Neurology. 2024 Oct 22;103(8):e209828. doi: 10.1212/WNL.0000000000209828. Epub 2024 Sep 16. PMID 39284112
- [Background] Cheng X, Su Y, Wang Q, Gao F, Ye X, Wang Y, Xia Y, Fu J, Shen Y, Al-Shahi Salman R, Dong Q. Neurofilament light chain predicts risk of recurrence in cerebral amyloid angiopathy-related intracerebral hemorrhage. Aging (Albany NY). 2020 Nov 18;12(23):23727-23738. doi: 10.18632/aging.103927. Epub 2020 Nov 18. PMID 33221749
- [Background] Wang SY, Chen W, Xu W, Li JQ, Hou XH, Ou YN, Yu JT, Tan L. Neurofilament Light Chain in Cerebrospinal Fluid and Blood as a Biomarker for Neurodegenerative Diseases: A Systematic Review and Meta-Analysis. J Alzheimers Dis. 2019;72(4):1353-1361. doi: 10.3233/JAD-190615. PMID 31744001
- [Background] Palmqvist S, Janelidze S, Stomrud E, Zetterberg H, Karl J, Zink K, Bittner T, Mattsson N, Eichenlaub U, Blennow K, Hansson O. Performance of Fully Automated Plasma Assays as Screening Tests for Alzheimer Disease-Related beta-Amyloid Status. JAMA Neurol. 2019 Sep 1;76(9):1060-1069. doi: 10.1001/jamaneurol.2019.1632. PMID 31233127
- [Background] Gatti L, Tinelli F, Scelzo E, Arioli F, Di Fede G, Obici L, Pantoni L, Giaccone G, Caroppo P, Parati EA, Bersano A. Understanding the Pathophysiology of Cerebral Amyloid Angiopathy. Int J Mol Sci. 2020 May 13;21(10):3435. doi: 10.3390/ijms21103435. PMID 32414028
- [Background] Greenberg SM, Bacskai BJ, Hernandez-Guillamon M, Pruzin J, Sperling R, van Veluw SJ. Cerebral amyloid angiopathy and Alzheimer disease - one peptide, two pathways. Nat Rev Neurol. 2020 Jan;16(1):30-42. doi: 10.1038/s41582-019-0281-2. Epub 2019 Dec 11. PMID 31827267
- [Background] Banerjee G, Ambler G, Keshavan A, Paterson RW, Foiani MS, Toombs J, Heslegrave A, Dickson JC, Fraioli F, Groves AM, Lunn MP, Fox NC, Zetterberg H, Schott JM, Werring DJ. Cerebrospinal Fluid Biomarkers in Cerebral Amyloid Angiopathy. J Alzheimers Dis. 2020;74(4):1189-1201. doi: 10.3233/JAD-191254. PMID 32176643
- [Background] Charidimou A, Boulouis G, Frosch MP, Baron JC, Pasi M, Albucher JF, Banerjee G, Barbato C, Bonneville F, Brandner S, Calviere L, Caparros F, Casolla B, Cordonnier C, Delisle MB, Deramecourt V, Dichgans M, Gokcal E, Herms J, Hernandez-Guillamon M, Jager HR, Jaunmuktane Z, Linn J, Martinez-Ramirez S, Martinez-Saez E, Mawrin C, Montaner J, Moulin S, Olivot JM, Piazza F, Puy L, Raposo N, Rodrigues MA, Roeber S, Romero JR, Samarasekera N, Schneider JA, Schreiber S, Schreiber F, Schwall C, Smith C, Szalardy L, Varlet P, Viguier A, Wardlaw JM, Warren A, Wollenweber FA, Zedde M, van Buchem MA, Gurol ME, Viswanathan A, Al-Shahi Salman R, Smith EE, Werring DJ, Greenberg SM. The Boston criteria version 2.0 for cerebral amyloid angiopathy: a multicentre, retrospective, MRI-neuropathology diagnostic accuracy study. Lancet Neurol. 2022 Aug;21(8):714-725. doi: 10.1016/S1474-4422(22)00208-3. PMID 35841910